CLINICAL TRIAL: NCT05629052
Title: TrEatment Approach in the Multimodal Era Registry
Acronym: TEAM
Status: Active, not recruiting | Type: Observational
Sponsor: International CTEPH Association (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: TEAM registry
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; CTEPH
Keywords: Chronic thromboembolic pulmonary hypertension; CTEPH; Pulmonary endarterectomy; PEA; Balloon pulmonary angioplasty; BPA; Multimodal treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Pulmonary endarterectomy — Surgical removal of a chronic clot from the pulmonary artery
  Other Names: PEA; Pulmonary thromboendarterectomy (PTE); PTE
Procedure: Balloon pulmonary angioplasty — Catheter-based intervention to dilate occluded pulmonary vessels through the insertion and inflation of a small balloon
  Other Names: BPA
Drug: Pulmonary hypertension (PH)-specific medication — Treatment with any PH-specific medication, i.e. endothelin receptor antagonists, phosphodiesterase type 5 inhibitors, soluble guanylate cyclase stimulators, drugs acting on the prostanoid pathway and prostaglandin I2 receptor agonists

SUMMARY:
The goal of this observational patient registry is to learn how expert centers treat patients with chronic thromboembolic pulmonary hypertension (CTEPH). CTEPH is a condition in which blood clots block the blood vessels in the lungs. There are currently three treatment options for patients with CTEPH:

* surgery to remove blood clots from large vessels in the lungs (pulmonary endarterectomy (PEA))
* the use of a small balloon to unblock smaller blood vessels (balloon pulmonary angioplasty (BPA))
* drugs

Patients can also receive a combination of these treatments.

The main question this registry aims to answer are:

* How many patients receive a given kind of treatment?
* How do expert centers combine the different treatments?
* Are patients doing better after they receive a given kind of treatment?
* How many patients are alive 1, 3 and 5 years after they receive a given kind of treatment?

Participants will receive the same treatments that they would receive if they did not participate in the study. During the study, patients will visit their doctors as they would do normally. The doctors will collect information on the patients' health and enter it into the study database. The follow-up time will be at least 3 years for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Newly referred patient with CTEPH or chronic thromboembolic pulmonary disease (CTEPD) without PH according to the following criteria:

   1. Mean pulmonary arterial pressure (mPAP) > 20 mmHg at rest with pulmonary vascular resistance (PVR) > 2 Wood units (WU); or if mPAP ≤ 20 mmHg or PVR ≤ 2 WU at rest, have exercise limitations from CTEPD without PH
   2. Abnormal ventilation perfusion scan, pulmonary angiogram, computer tomographic pulmonary angiogram, or magnetic resonance pulmonary angiogram confirming CTEPD as recommended by standard guidelines
2. Treatment with anticoagulation for ≥ 3 months before diagnosis of CTEPH or CTEPD without PH
3. Naïve to interventional treatment (both PEA and BPA)
4. Pre-treatment with PH-specific medication for ≤ 12 months, or no medical pre-treatment, at enrollment
5. Willing and able to provide informed consent in order to participate in the study (informed consent signed)
6. Age ≥ 18 years
7. CTEPH-specific treatment must be modified or initiated at the participating site

Exclusion Criteria:

1. Main cause of PH other than CTEPH
2. Participating in an interventional clinical trial at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from CTEPH or CTEPD without PH who are newly referred to an expert center and who meet all of the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Utilization and combination of treatment modalities | Min. 3 years
  Proportion of patients undergoing a certain type of treatment modality, or a certain combination of modalities
3-year survival | 3 years after last intervention
  Proportion of patients alive 3 years after the last intervention recorded in the registry, or after start of medical treatment for patients not undergoing any interventional treatment

SECONDARY OUTCOMES:
Complications of treatment interventions (per patient) | Min. 3 years
  Proportion of patients experiencing complications from BPA or PEA
Complications of treatment interventions (per BPA session) | Min. 3 years
  Proportion of BPA sessions associated with complications
1-year survival | 1 year after last intervention
  Proportion of patients alive 1 year after the last intervention recorded in the registry, or after start of medical treatment for patients not undergoing any interventional treatment
5-year survival | 5 year after last intervention
  Proportion of patients alive 5 years after the last intervention recorded in the registry, or after start of medical treatment for patients not undergoing any interventional treatment
Changes in PH-specific medication | Min. 3 years
  Proportion of patients experiencing a change in PH-specific medication during the study
Reason why PEA was not performed | Min. 3 years
  The main reason why PEA was not performed as chosen by the investigator from a list of pre-defined reasons
Reason why BPA was not performed | Min. 3 years
  The main reason why BPA was not performed as chosen by the investigator from a list of pre-defined reasons

OTHER OUTCOMES:
Number of unplanned hospitalizations | Min. 3 years
  Proportion of patients experiencing an unplanned hospitalization (i.e. not considering planned hospitalizations for study procedures such as PEA or BPA)
Timing of unplanned hospitalizations | Min. 3 years
  Analysis of the timing of unplanned hospitalization for patients experiencing an unplanned hospitalization (i.e. not considering planned hospitalizations for study procedures such as PEA or BPA)
Frequency of QoL assessment | Min. 3 years
  Proportion of patients undergoing QoL assessment by means of a validated questionnaire during the study
Type of QoL questionnaire | Min. 3 years
  Proportion of patients undergoing QoL assessment using a certain validated questionnaire during the study

CONTACTS AND LOCATIONS:
Overall Officials: Nick H Kim, MD, Principal Investigator — University of California, San Diego
Locations (25):
- United States (4):
  - University of California San Diego, San Diego, California
  - Northwestern University, Evanston, Illinois
  - Duke University, Durham, North Carolina
  - UT Southwestern, Dallas, Texas
- Hospital Universitario Fundación Favaloro, Buenos Aires, Argentina
- University Hospital Vienna, Vienna, Austria
- University Hospitals Leuven, Leuven, Belgium
- Santa Casa, Porto Alegre, Brazil
- Toronto General Hospital, Toronto, Ontario, Canada
- China-Japan Friendship Hospital, Beijing, China
- Shaio Clinic Foundation, Bogotá, Colombia
- General University Hospital, Prague, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- Kerckhoff Clinic, Department of Thoracic Surgery, Bad Nauheim, Germany
- Narayana Institute of Cardiac Science, Bangalore, India
- University of Bologna, Bologna, Italy
- Japan (2):
  - Okayama Medical Center, Okayama
  - National Cerebral and Cardiovascular Center, Osaka
- National Heart Institute, Mexico City, Mexico
- Poland (2):
  - Department of Cardiac and Vascular Diseases, John Paul II Hospital, Krakow
  - Department of Pulmonary Circulation, Thromboembolic Diseases and Cardiology, European Health Center Otwock, Otwock
- National Heart Centre of Singapore, Singapore, Singapore
- Pulmonary Hypertension Unit, Hospital 12 de Octubre, Madrid, Spain
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)
- Royal Papworth Hospital, Cambridge, United Kingdom

REFERENCES:
- See also: Description of the registry on the website of the International CTEPH Association — https://www.cteph-association.org/team-registry.html